CLINICAL TRIAL: NCT04710862
Title: The Effects of Respiratory-Based Treatment for Muscle Tension Dysphonia: A Randomized Controlled Trial
Brief Title: The Effects of Respiratory Training on Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, Soren Lowell, Professor, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-132
Record Dates: First submitted 2020-11-30; First posted 2021-01-15 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Muscle Tension Dysphonia
Keywords: voice; voice disorder; treatment; respiratory; muscle tension dysphonia; training
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing training with a device (Sham Training as Control) (Active Comparator): Respiratory intervention delivered once a week for 6 weeks, after two initial baseline testing sessions. Participants will perform exhalation exercises through a breathing device. Homework activities will be assigned. Post-training testing sessions will also be conducted.
  Interventions: Behavioral: Breathing training with a device
- Breathing training without a device (Respiratory Lung Volume Training) (Active Comparator): Respiratory intervention delivered once a week for 6 weeks, after two initial baseline testing sessions. Participants will receive training on the use of breathing techniques without a device, but with visual feedback throughout training. Homework activities will be assigned. Post-training testing sessions will also be conducted.
  Interventions: Behavioral: Breathing training without a device

INTERVENTIONS:
Behavioral: Breathing training without a device — Breathing training without a mouth device
  Arms: Breathing training without a device (Respiratory Lung Volume Training)
Behavioral: Breathing training with a device — Breathing training with a mouth device
  Arms: Breathing training with a device (Sham Training as Control)

SUMMARY:
Primary muscle tension dysphonia is a voice disorder that involves excessive and poorly coordinated muscle activity affecting multiple subsystems that are involved in speech production, in the absence of structural or neurologic abnormalities of the larynx. Primary muscle tension dysphonia (MTD) is one of the most common forms of voice disorders, accounting for at least 40% of patients seen in voice clinics. Perceptually the voice sounds hoarse and strained, with reduced loudness and pitch range, and people with MTD find speaking very effortful and fatiguing. The physiological abnormalities that characterize MTD are considered multifactorial, and include over-activity of muscles in and around the larynx, laryngeal constriction patterns, and abnormal speech breathing patterns. However, standard treatment approaches for MTD primarily address laryngeal function, including repositioning of laryngeal structures, reducing activity in the intrinsic and extrinsic laryngeal muscles, and altering vibratory patterns. Although voice improvement may follow these treatments, many people with MTD show recurrence of voice problems after only a few months, and some do not improve with treatment. These findings highlight the need for alternative treatments that address the respiratory contributions to MTD, which directly affect the phonatory system. The goal of this project is to compare the effects of two respiratory-based training conditions in people with MTD. A randomized group design will be implemented to determine the respiratory and acoustic effects of each condition. We will determine the effects of each condition immediately after and then 3 and 6 months after training completion to assess short- and long-term training effects. We propose that respiratory training will have a positive effect on related laryngeal behavior and voice. The proposed project has the potential to substantially advance the evidence-based treatment options for MTD, providing a vital step toward reducing the debilitating effects of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Self-report of general good health other than voice disorder
* Self-report of normal pulmonary function
* Non-smoker status for at least the last 5 years
* English as their primary language to avoid potential linguistically-based differences in acoustic measures of voice
* Adequate visual acuity (with or without corrective lenses) to read basic graphs and print, as determined with visual screening
* No evidence of current organic or neurologic laryngeal pathology, as assessed by nasolaryngoscopy examination and reviewed by a laryngologist
* No prior surgery to the vocal folds
* Do not report difficulty with swallowing
* Not currently receiving voice therapy or other voice treatment that cannot be discontinued
* Do not report a bilateral, severe to profound hearing loss
* Willingness to be recorded for data collection that is necessary for this study
* Have a confirming diagnosis of Muscle Tension Dysphonia from an otolaryngologist and speech-language pathologist
* Demonstrate quantified auditory-perceptual dysphonia and acoustic dysphonia (Cepstral/Spectral Index of Dysphonia) that exceed normative values for the participant's age and sex
* Based on the nasolaryngoscopy examination and assessment performed by the otolaryngologist, show one or more patterns of supraglottic activity that are consistent with adducted vocal fold hyperfunction
* Show no evidence of abnormal, incomplete vocal fold closure patterns as determined on the videostroboscopy assessment (patterns of posterior glottal gaps are normal and expected)
* Show no evidence of additional neurological voice disorders such as spasmodic dysphonia or vocal fold paralysis
* Show elevated hyolaryngeal position that exceeds normative expectations as determined through quantitative analysis of ultrasonographic laryngeal images measuring change from rest to phonation
* Demonstrate voice problems that have persisted for ≥2 months
* Demonstrate self-reported increase in speaking effort
* Show evidence of speech breathing abnormalities relative to accepted normative values

Exclusion Criteria:

* Ages 17 or younger
* Self-report of major health problems
* Self-report of pulmonary disease such as asthma, chronic obstructive pulmonary disease, or emphysema
* Current smoker status or prior smoker status within the last 5 years
* English not the primary language
* Inadequate visual acuity (with corrective lenses if applicable) to read basic graphs and print as determined by failing a visual screening
* Evidence of current organic or neurologic laryngeal pathology, as assessed by nasolaryngoscopy examination and reviewed by a laryngologist
* Prior surgery to the vocal folds
* Currently receiving voice therapy or other voice treatment that cannot be discontinued
* Self-report of a bilateral, severe to profound hearing loss
* Not willing to be recorded for data collection that is necessary for this study
* No confirming diagnosis of Muscle Tension Dysphonia from an otolaryngologist and speech-language pathologist
* Do not demonstrate quantified auditory-perceptual dysphonia and acoustic dysphonia (Cepstral/Spectral Index of Dysphonia) that exceed normative values for the participant's age and sex
* Based on the nasolaryngoscopy examination and assessment performed by the otolaryngologist, do not show one or more patterns of supraglottic activity that are consistent with adducted vocal fold hyperfunction
* Show evidence of abnormal, incomplete vocal fold closure patterns as determined on the videostroboscopy assessment (patterns of posterior glottal gaps are normal and expected)
* Show evidence of additional neurological voice disorders such as spasmodic dysphonia or vocal fold paralysis
* Do not show elevated hyolaryngeal position that exceeds normative expectations as determined through quantitative analysis of ultrasonographic laryngeal images measuring change from rest to phonation
* Demonstrate voice problems that have persisted for less than 2 months
* Do not demonstrate self-reported increase in speaking effort
* Do not show evidence of speech breathing abnormalities relative to accepted normative values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soren Y Lowell, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants were enrolled in the study. After initial testing to determine inclusion and exclusion criteria, 3 participants were excluded due to not meeting all inclusion/exclusion criteria. The remaining 24 participants were randomized into the two intervention groups, 12 per group.
Groups:
- Breathing Training Without a Device: Respiratory intervention delivered once a week for 6 weeks, after two initial baseline testing sessions. Participants will receive training on the use of breathing techniques without a device, but with visual feedback throughout training. Homework activities will be assigned. Post-training testing sessions will also be conducted.
  Breathing training without a device: Breathing training without a mouth device
Period: Overall Study
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device
Started | 12 | 12
Completed | 12 (Number of participants who completed study endpoints for primary intervention phase) | 12 (Number of participants who completed study endpoints for primary intervention phase)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (15.4) | 55.4 (12.6) | 58.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Lung Volume Initiation - Relative to Resting Expiratory Level [Mean (Standard Deviation); unit: % vital capacity relative to rest level] | 19.01 (6.11) | 15.05 (7.00) | 17.03 (6.56)
Lung Volume Termination - Relative to Resting Expiratory Level [Mean (Standard Deviation); unit: % vital capacity relative to rest level] | -1.07 (4.40) | -4.55 (5.38) | -2.81 (4.89)
Lung Volume Excursion [Mean (Standard Deviation); unit: % vital capacity relative to rest level] | 20.08 (4.94) | 19.60 (8.04) | 19.84 (6.49)
% Vital Capacity per Syllable [Mean (Standard Deviation); unit: % vital capacity relative to rest level] | 1.42 (0.48) | 1.44 (0.65) | 1.43 (0.57)
Cepstral/Spectral Index of Dysphonia [Mean (Standard Deviation); unit: units on a scale] — The Cepstral/Spectral Index of Dysphonia is a multivariate measure that indicates the acoustic severity of voice, and is calculated from the recorded acoustic voice signal. The scale generally ranges from 0 to 100, although negative values and values greater than 100 are possible. A score of zero or a low score indicates no acoustic dysphonia (no voice abnormality) or little dysphonia, whereas a high score or score of 100 indicates high severity or maximal severity of acoustic dysphonia.
  units on a scale | 30.73 (13.18) | 29.59 (8.43) | 30.16 (10.81)
Cepstral Peak Prominence [Mean (Standard Deviation); unit: decibels (dB)] — The Cepstral Peak Prominence measure indicates the regularity, or periodicity, of the voice, and is calculated from the recorded acoustic voice signal. A low score such as 2.0 indicates lower regularity in the voice, or greater severity of voice disturbance, whereas a higher score indicates greater regularity in the voice, or less severity of voice disturbance. The values of this measure can theoretically range from zero to any positive integer value.
  decibels (dB) | 4.96 (1.24) | 4.85 (0.96) | 4.91 (1.10)
Auditory-Perceptual Overall Voice Severity [Mean (Standard Deviation); unit: units on a scale] — Auditory-Perceptual Overall Voice Severity is a measure that indicates the perceptual severity of the voice, and is determined by listeners who rate the overall severity of how the voice sounds on a Visual Analog Scale that ranges from 0 to 100. A score of zero or a low score indicates no or little perceived dysphonia (voice abnormality), whereas a high score or score of 100 indicates high or maximal perceived severity of dysphonia.
  units on a scale | 35.16 (24.40) | 30.85 (20.71) | 33.01 (22.56)
Speaking Effort [Mean (Standard Deviation); unit: units on a scale] — Speaking effort is a self-rated measure that indicates how much effort the participant feels while speaking, and is rated on a Visual Analog Scale from 0 (no effort) to 100 (maximal effort). This measure represents the difference of what the participant feels is their typical amount of speaking effort minus their rating of comfortable speaking effort. The range of this difference score is usually between 0 to 100. A low score indicates that the participant feels low amounts of effort while speaking, whereas a high score indicates that a participant feels speaking is very effortful.
  units on a scale | 56.56 (22.43) | 58.46 (13.99) | 57.51 (18.21)
Voice Handicap Index-10 [Mean (Standard Deviation); unit: units on a scale] — The Voice Handicap Index-10 is a questionnaire in which the participant rates the amount of handicap they feel from their voice disorder. Each of 10 questions is rated between a score of 0 (no handicap) to 4 (extreme handicap). Total scores on this questionnaire can range between 0 to 40, with a low score indicating that the participant feels low amounts of handicap or life impact from their voice disorder, whereas a high score indicates that a participant feels high amounts of handicap from their voice disorder.
  units on a scale | 19.96 (6.49) | 19.75 (9.33) | 19.86 (7.91)

OUTCOME MEASURES:

1. Primary Outcome: Post Training Lung Volume Initiation
Description: Average level of lung volume at which speech breaths are initiated, expressed in percent vital capacity relative to resting expiratory level.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: % vital capacity relative to rest level
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
% vital capacity relative to rest level | 21.07 (4.94) | 27.04 (7.71)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p < 0.0005, Mixed Models Analysis

2. Primary Outcome: Post Training Lung Volume Termination
Description: Average level of lung volume at which speech breaths are terminated, expressed in percent vital capacity relative to resting expiratory level.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: % vital capacity relative to rest level
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
% vital capacity relative to rest level | -0.44 (5.26) | 2.29 (5.04)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p < 0.0005, Mixed Models Analysis

3. Primary Outcome: Post Training Lung Volume Excursion
Description: Average level of lung volume at which speech breaths are terminated, expressed in percent vital capacity.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: % vital capacity
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
% vital capacity | 21.51 (4.81) | 24.74 (6.48)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p = 0.012, Mixed Models Analysis

4. Primary Outcome: Post Training Cepstral Peak Prominence
Description: Average energy in first cepstral peak relative to overall cepstral energy, measured in cepstral decibels. The Cepstral Peak Prominence measure indicates the regularity, or periodicity, of the voice, and is calculated from the recorded acoustic voice signal. A low score such as 2.0 indicates lower regularity in the voice, or greater severity of voice disturbance, whereas a higher score indicates greater regularity in the voice, or less severity of voice disturbance. The values of this measure can theoretically range from zero to any positive integer value.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
decibels (dB) | 4.86 (1.10) | 5.31 (0.81)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p = 0.001, Mixed Models Analysis

5. Primary Outcome: Post Training Cepstral/Spectral Index of Dysphonia
Description: The Cepstral/Spectral Index of Dysphonia is a multivariate measure that indicates the acoustic severity of voice, and is calculated from the recorded acoustic voice signal. The scale generally ranges from 0 to 100, although negative values and values greater than 100 are possible. A score of zero or a low score indicates no acoustic dysphonia (no voice abnormality) or little dysphonia, whereas a high score or score of 100 indicates high severity or maximal severity of acoustic dysphonia.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
units on a scale | 29.03 (14.06) | 21.96 (9.76)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p = 0.004, Mixed Models Analysis

6. Secondary Outcome: Post Training Auditory-Perceptual Overall Severity of Voice Disorder
Description: Auditory-Perceptual Overall Voice Severity is a measure that indicates the perceptual severity of the voice, and is determined by listeners who rate the overall severity of how the voice sounds on a Visual Analog Scale that ranges from 0 to 100. A score of zero or a low score indicates no or little perceived dysphonia (voice abnormality), whereas a high score or score of 100 indicates high or maximal perceived severity of dysphonia.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
units on a scale | 33.29 (24.18) | 18.78 (12.28)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p = 0.001, Mixed Models Analysis

7. Secondary Outcome: Post Training Voice Handicap Index-10
Description: The Voice Handicap Index-10 is a questionnaire in which the participant rates the amount of handicap they feel from their voice disorder. Each of 10 questions is rated between a score of 0 (no handicap) to 4 (extreme handicap). Total scores on this questionnaire can range between 0 to 40, with a low score indicating that the participant feels low amounts of handicap or life impact from their voice disorder, whereas a high score indicates that a participant feels high amounts of handicap from their voice disorder.
Time Frame: Assessed after completion of 6-week training period, approximately 7 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
Number analyzed (Participants) | 12 | 12
units on a scale | 14.38 (6.63) | 12.13 (6.02)
Statistical Analysis 1: Comparison: Breathing Training With a Device (Sham Training as Control) vs Breathing Training Without a Device (Respiratory Lung Volume Training); Test type: Superiority; p = 0.328, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the period in which each participant completed baseline testing, training, and post-testing, or 8 weeks total.
Arm/Group | Breathing Training With a Device (Sham Training as Control) | Breathing Training Without a Device (Respiratory Lung Volume Training)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04710862/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04710862/SAP_001.pdf